CLINICAL TRIAL: NCT04071353
Title: Observational Cohort Study of Clinical Outcomes After Antiviral Therapy in Chronic Hepatitis C Patients
Brief Title: Observational Cohort Study of Clinical Outcomes After Antiviral Therapy for Chronic Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of liver disease, Beijing Ditan Hospital
Other Study IDs: DTXY021
Record Dates: First submitted 2019-08-18; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; Interferon; Ribavirin; Clinical outcome
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Interferons; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interferon combined with ribavirin group: Interferon combined with ribavirin (PR) antiviral therapy (PR treatment for 6 months or more) in patients with chronic hepatitis C, collect basic data before antiviral therapy, and during the PR antiretroviral treatment period, Follow-up was performed every 3-6 months in March, June, September, December, DAAs antiviral treatment during January, March, and withdrawal follow-up, and clinical biochemistry, HCV RNA, and serological markers were used during follow-up ( anti-HCV), AFP and liver imaging (liver ultrasound) examination.
  Interventions: Drug: Interferon; Drug: ribavirin
- DAAs treatment group: Patients with chronic hepatitis C treated with direct acting antivirals (DAAs), collect basic data before antiviral therapy, and during the period of PR antiviral treatment, January, March, June, September, December Follow-up was performed every 3-6 months during January, March, and withdrawal follow-up during DAAs antiviral therapy. Clinical biochemistry, HCV RNA and serological markers (anti-HCV), AFP, and liver imaging were performed at follow-up. Liver ultrasound) check.
  Interventions: Drug: DAAs

INTERVENTIONS:
Drug: Interferon — Interferon combined with ribavirin antiviral therapy
  Groups: Interferon combined with ribavirin group
Drug: ribavirin — Interferon combined with ribavirin antiviral therapy
  Groups: Interferon combined with ribavirin group
Drug: DAAs — DAAs antiviral treatment
  Groups: DAAs treatment group

SUMMARY:
This study was a clinical observational cohort study of two-way, non-intervention long-term dynamic follow-up. Enrolled in the Department of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, with interferon combined with ribavirin (PR) antiviral therapy (PR treatment greater than or equal to 6 months) and/or direct acting antivirals (DAAs) In patients with chronic hepatitis C, the baseline, antiviral treatment and withdrawal follow-up data before the antiviral treatment were collected, and the patients were followed up for 3-6 months. Clinical data such as clinical biochemistry, HCV RNA and serological markers (anti-HCV), AFP and liver imaging (liver ultrasound) were collected during the study period. At least 144 weeks of observation on the virological response and clinical outcome of anti-viral treatment of chronic hepatitis C, the main evaluation index of liver cancer and decompensated liver cirrhosis after stopping the drug, and exploring the antiviral treatment of patients Long-term virological response and clinical outcomes, clarifying their influencing factors.

DETAILED DESCRIPTION:
This study was a clinical observational cohort study of two-way, non-intervention long-term dynamic follow-up. Enrolled in the Department of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, with interferon combined with ribavirin (PR) antiviral therapy (PR treatment greater than or equal to 6 months) and/or direct acting antivirals (DAAs) In patients with chronic hepatitis C, the baseline, antiviral treatment and withdrawal follow-up data before the antiviral treatment were collected, and the patients were followed up for 3-6 months. Clinical data such as clinical biochemistry, HCV RNA and serological markers (anti-HCV), AFP and liver imaging (liver ultrasound) were collected during the study period. At least 144 weeks of observation on the virological response and clinical outcome of anti-viral treatment of chronic hepatitis C, the main evaluation index of liver cancer and decompensated liver cirrhosis after stopping the drug, and exploring the antiviral treatment of patients Long-term virological response and clinical outcomes, clarifying their influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C patients treated with interferon plus ribavirin (PR) antiviral therapy (PR treatment greater than or equal to 6 months) and/or direct antiviral drugs (DAAs)

Exclusion Criteria:

* Co-infected with hepatitis B virus or human immunodeficiency virus
* Had an autoimmune disease, liver tumour, or severe cardiac disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients treated with interferon plus ribavirin (PR) antiviral therapy (PR treatment greater than or equal to 6 months) and/or direct antiviral drugs (DAAs). All patients with chronic hepatitis C were eligible for the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis C (2015).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of liver cancer | up to 144 weeks
  The incidence of liver cancer after anti-viral treatment of chronic hepatitis C
The incidence of decompensated cirrhosis | up to 144 weeks
  The incidence of decompensated cirrhosis after anti-viral treatment of chronic hepatitis C

SECONDARY OUTCOMES:
Percentage of persistent virological response or relapse | up to 144 weeks
  Percentage of persistent virological response or relapse after antiviral therapy for chronic hepatitis C
Related factors of liver cancer | up to 144 weeks
  Related factors including viral indicators (HCV RNA content, anti-HCV), clinical biochemical indicators (ALT, AST, ALB, Tbil), blood routine and coagulation function indicators (PTA) and serum AFP and liver ultrasound results of liver cancer after anti-viral treatment of chronic hepatitis C
Related factors of decompensated cirrhosis | up to 144 weeks
  Related factors including viral indicators (HCV RNA content, anti-HCV), clinical biochemical indicators (ALT, AST, ALB, Tbil), blood routine and coagulation function indicators (PTA) and serum AFP and liver ultrasound results of decompensated cirrhosis after anti-viral treatment of chronic hepatitis C

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, phD/MD, Study Director — Beijing Ditan Hospital
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China